CLINICAL TRIAL: NCT04343651
Title: A Phase 2, Randomized, Double Blind, Placebo Controlled Study to Evaluate the Efficacy and Safety of Leronlimab for Mild to Moderate Coronavirus Disease 2019 (COVID-19)
Brief Title: Study to Evaluate the Efficacy and Safety of Leronlimab for Mild to Moderate COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CytoDyn, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CD10_COVID-19
Record Dates: First submitted 2020-03-31; First posted 2020-04-13 (Actual); Results first posted 2023-01-04 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2022-12

CONDITIONS: Coronavirus Disease 2019
Keywords: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — leronlimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): The placebo comparator consists of the formulation buffer for leronlimab, i.e., the placebo is the same as the active arm without leronimab. The placebo is presented in the same container closure at the same fill volume as the active (nominal 1mL fill volume). The formulation buffer contains histidine, glycine, sodium chloride, sorbitol, polysorbate 20 and sterile water for injections.
  Interventions: Drug: Placebo
- 700mg Leronlimab (Experimental): Each vial of active contains 175mg of leronlimab at a concentration of 175mg/ml (nominal 1mL fill volume) in formulation buffer containing histidine, glycine, sodium chloride, sorbitol, polysorbate 20 and sterile water for injections.
  Interventions: Drug: Leronlimab (700mg)

INTERVENTIONS:
Drug: Placebo — Placebo
  Arms: Placebo
Drug: Leronlimab (700mg) — Leronlimab (PRO) 140 is a humanized IgG4, monoclonal antibody (mAb) to the C-C chemokine receptor type 5 (CCR5)
  Other Names: PRO 140
  Arms: 700mg Leronlimab

SUMMARY:
This is a Phase 2, two-arm, randomized, double blind, placebo controlled multicenter study to evaluate the safety and efficacy of leronlimab (PRO 140) in patients with mild-to-moderate symptoms of respiratory illness caused by coronavirus 2019 infection.

DETAILED DESCRIPTION:
This is a Phase 2, two-arm, randomized, double blind, placebo controlled multicenter study to evaluate the safety and efficacy of leronlimab (PRO 140) in patients with mild-to-moderate symptoms of respiratory illness caused by coronavirus 2019 infection. Patients will be randomized to receive weekly doses of 700 mg leronlimab (PRO 140), or placebo. Leronlimab (PRO 140) and placebo will be administered via subcutaneous injection.

The study will have three phases: Screening Period, Treatment Period, and Follow-Up Period.

A total of 75 subjects will be randomized 2:1 in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adult ≥ 18 years of age at time of enrollment.
2. Subjects with mild-to-moderate symptoms of respiratory illness caused by coronavirus 2019 infection as defined below:

   Mild (uncomplicated) Illness:
   * Diagnosed with COVID-19 by a standardized RT-PCR assay AND
   * Mild symptoms, such as fever, rhinorrhea, mild cough, sore throat, malaise, headache, muscle pain, or malaise, but with no shortness of breath AND
   * No signs of a more serious lower airway disease AND
   * RR<20, HR <90, oxygen saturation (pulse oximetry) > 93% on room air

   Moderate Illness:
   * Diagnosed with COVID-19 by a standardized RT-PCR assay AND
   * In addition to symptoms above, more significant lower respiratory symptoms, including shortness of breath (at rest or with exertion) OR
   * Signs of moderate pneumonia, including RR ≥ 20 but <30, HR ≥ 90 but less than 125, oxygen saturation (pulse oximetry) > 93% on room air AND
   * If available, lung infiltrates based on X-ray or CT scan < 50% present
3. Clinically normal resting 12-lead ECG at Screening Visit or, if abnormal, considered not clinically significant by the Principal Investigator.
4. Subject (or legally authorized representative) provides written informed consent prior to initiation of any study procedures.
5. Understands and agrees to comply with planned study procedures.
6. Women of childbearing potential must agree to use at least one medically accepted method of contraception (e.g., barrier contraceptives [condom, or diaphragm with a spermicidal gel], hormonal contraceptives [implants, injectables, combination oral contraceptives, transdermal patches, or contraceptive rings], or intrauterine devices) for the duration of the study.

Exclusion Criteria:

1. Subjects showing signs of acute respiratory distress syndrome (ARDS) or respiratory failure necessitating mechanical ventilation at the time of screening;
2. History of severe chronic respiratory disease and requirement for long-term oxygen therapy;
3. Subjects showing signs of clinical jaundice at the time of screening;
4. History of moderate and severe liver disease (Child-Pugh score >12);
5. Subjects requiring Renal Replacement Therapy (RRT) at the time of screening;
6. History of severe chronic kidney disease or requiring dialysis;
7. Any uncontrolled active systemic infection requiring admission to an intensive care unit (ICU); Note: Subjects infected with chronic hepatitis B virus or hepatitis C virus will be eligible for the study if they have no signs of hepatic decompensation.

   Note: Subjects infected with HIV-1 will be eligible for the study with undetectable viral load and are on a stable ART regimen. Investigators are required to review the subjects' medical records to confirm HIV-1 RNA suppression within the previous 3 months.

   Note: Empirical antibiotic treatment for secondary bacterial infections is allowed during the course of study.
8. Patients with malignant tumor, or other serious systemic diseases;
9. Patients who are participating in other clinical trials;
10. Patients who have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to leronlimab (PRO 140) are not eligible; and
11. Inability to provide informed consent or to comply with test requirements

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-07-21 (Actual); Study Completion 2021-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angela Ritter, MD, Principal Investigator — Center for Advanced Research and Education
Locations (12):
- United States (12):
  - University of California, Los Angeles, Los Angeles, California
  - Palmtree Clinical Research, Inc., Palm Springs, California
  - Eisenhower Health, Rancho Mirage, California
  - Yale, New Haven, Connecticut
  - Center for Advanced Research & Education (CARE), Gainesville, Georgia
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Atlantic Health System Hospital, Morristown, New Jersey
  - Montefiore Medical Center, The Bronx, New York
  - White Plains Hospital, White Plains, New York
  - Novant Health, Charlotte, North Carolina
  - Ohio Health, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Seethamraju H, Yang OO, Loftus R, Ogbuagu O, Sammartino D, Mansour A, Sacha JB, Ojha S, Hansen SG, Arman AC, Lalezari JP. A Randomized Placebo-Controlled Trial of Leronlimab in Mild-To-Moderate COVID-19. Clin Ther. 2024 Nov;46(11):891-899. doi: 10.1016/j.clinthera.2024.08.019. Epub 2024 Sep 30. PMID 39353749
- See also: NEWS2 Score — https://www.rcplondon.ac.uk/projects/outputs/national-early-warning-score-news-2

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States. The first participant was randomized on 30-Apr-2020. Data submitted represent analysis performed on data collected after all patients completed the Follow UP period.
Pre-assignment Details: 126 patients were screened, 40 were screen failures.
Groups:
- Placebo: Placebos: Placebo
  Patients who meet the below criteria will be randomized 2:1 to receive weekly doses of 700 mg leronlimab (PRO 140), or placebo. Leronlimab (PRO 140) and placebo will be administered via subcutaneous injection.
  Male or female adult ≥ 18 years of age at time of enrollment with mild-to-moderate symptoms of respiratory illness caused by coronavirus 2019 infection as defined below:
  Mild (uncomplicated) Illness:
  * Diagnosed with COVID-19 by a standardized RT-PCR assay AND
  * Mild symptoms, such as fever, rhinorrhea, mild cough, sore throat, malaise, headache, muscle pain, or malaise, but with no shortness of breath AND
  * No signs of a more serious lower airway disease AND
  * RR<20, HR <90, oxygen saturation (pulse oximetry) > 93% on room air
  Moderate Illness:
  * Diagnosed with COVID-19 by a standardized RT-PCR assay AND
  * In addition to symptoms above, more significant lower respiratory symptoms, including shortness of breath (at rest or with exertion) OR
  * Signs of moderate pneumonia, including RR ≥ 20 but <30, HR ≥ 90 but less than 125, oxygen saturation (pulse oximetry) > 93% on room air AND
  * If available, lung infiltrates based on X-ray or CT scan < 50% present
  Clinically normal resting 12-lead ECG at Screening Visit or, if abnormal, considered not clinically significant by the Principal Investigator.
- 700mg Leronlimab: Leronlimab (700mg): Leronlimab (PRO) 140 is a humanized IgG4, monoclonal antibody (mAb) to the C-C chemokine receptor type 5 (CCR5)
  Patients who meet the below criteria will be randomized 2:1 to receive weekly doses of 700 mg leronlimab (PRO 140), or placebo. Leronlimab (PRO 140) and placebo will be administered via subcutaneous injection.
  Male or female adult ≥ 18 years of age at time of enrollment with mild-to-moderate symptoms of respiratory illness caused by coronavirus 2019 infection as defined below:
  Mild (uncomplicated) Illness:
  * Diagnosed with COVID-19 by a standardized RT-PCR assay AND
  * Mild symptoms, such as fever, rhinorrhea, mild cough, sore throat, malaise, headache, muscle pain, or malaise, but with no shortness of breath AND
  * No signs of a more serious lower airway disease AND
  * RR<20, HR <90, oxygen saturation (pulse oximetry) > 93% on room air
  Moderate Illness:
  * Diagnosed with COVID-19 by a standardized RT-PCR assay AND
  * In addition to symptoms above, more significant lower respiratory symptoms, including shortness of breath (at rest or with exertion) OR
  * Signs of moderate pneumonia, including RR ≥ 20 but <30, HR ≥ 90 but less than 125, oxygen saturation (pulse oximetry) > 93% on room air AND
  * If available, lung infiltrates based on X-ray or CT scan < 50% present
  Clinically normal resting 12-lead ECG at Screening Visit or, if abnormal, considered not clinically significant by the Principal Investigator.
Period: Overall Study
Arm/Group | Placebo | 700mg Leronlimab
Started | 29 | 57
Completed | 17 | 33
Not Completed | 12 | 24
Not completed — Physician Decision | 2 | 1
Not completed — Lost to Follow-up | 2 | 1
Not completed — Protocol Violation | 4 | 6
Not completed — Missing | 3 | 9
Not completed — Withdrawal by Subject | 0 | 4
Not completed — Death | 0 | 1
Not completed — Did not start treatment | 1 | 1
Not completed — Patient did not complete visits 3-6 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Modified Intent-to-Treat (mITT) population is defined as the set of subjects who have received at least one dose of leronlimab or placebo and is population used for the analysis of efficacy parameters or measurements.
  The Safety Population includes all subjects who received at least one dose of leronlimab or placebo. This population was used for the analysis of safety parameters or measurements. There were 84 subjects in the MITT and Safety Population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 700mg Leronlimab | Total
Number analyzed (Participants) | 28 | 56 | 84
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 42 | 63
  >=65 years | 7 | 14 | 21
Age, Continuous [Mean (Full Range); unit: years] | 55.36 [23 to 84] | 54.59 [30 to 79] | 54.85 [23 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 32 | 51
  Male | 9 | 24 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 18 | 28
  Not Hispanic or Latino | 17 | 35 | 52
  Unknown or Not Reported | 1 | 3 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 18 | 28
  Not Hispanic or Latino | 17 | 35 | 52
  Unknown or Not Reported | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 28 | 56 | 84
COVID SYMPTOMS SCORE [Count of Participants; unit: Participants] — Baseline symptoms assessed were fever, myalgia, dyspnea, and cough. Each symptom was graded from 0 to 3 [0=none, 1=mild, 2=moderate, and 3=severe]. The total score is calculated by summing all scores, with a higher score indicating a worse health state.
  The total score per patient ranged from 0 to 12 points.
  Participants
    Baseline symptom score less than or equal to 4 | 16 | 29 | 45
    Baseline symptom score greater than 4 | 12 | 27 | 39

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Total Symptom Score
Description: Clinical Improvement as assessed by change in total symptom score (for fever, myalgia, dyspnea and cough) by count of patients showing improvement, no change or worsened.
  Note: The total score per patient ranges from 0 to 12 points. Each symptom is graded from 0 to 3. [0=none, 1=mild, 2=moderate, and 3=severe]. Higher scores mean a worse outcome. A negative change from baseline shows an improvement in symptom score.
Time Frame: Clinical Improvement will be assessed at baseline and at EOT (day 14).
Population: The Modified Intent-to-Treat (mITT) population was defined as the set of subjects who received at least one dose of leronlimab (PRO 140) or placebo. This population was to be used for the analysis of efficacy parameters or measurements. At the time of this report, there were 84 subjects in the mITT population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | 700mg Leronlimab
Number analyzed (Participants) | 28 | 56
units on a scale | -3.4 (3.19) | -3.5 (3.03)
Statistical Analysis 1: Comparison: Placebo vs 700mg Leronlimab; Test type: Superiority; p = 0.818, ANCOVA

2. Secondary Outcome: Time to Clinical Resolution (TTCR)
Description: Defined as the time from initiation of study treatment to the resolution of clinical symptoms (fever, myalgia, dyspnea, cough).
  Data presented how the number of days at which a certain percentage of patients achieve resolution of symptoms, i.e., 50% of patients on placebo saw resolution of symptoms in 15 days, and 15 days for patients on leronlimab.
  The hazard ratio was 0.781, 95% Confidence Interval 0.43, 1.41 and the p-value was 0.4138.
  TTCR is defined as the duration from date of first exposure to treatment to the first occurrence of total symptom score equals 0.
Time Frame: Time (in days) from initiation of study treatment until resolution of clinical symptoms (fever, myalgia, dyspnea and cough).
Population: MITT
Measure: Number; unit: days
Arm/Group | Placebo | 700mg Leronlimab
Number analyzed (Participants) | 28 | 56
days
  25% subjects | 5 | 8
  50% subjects | 15 | 15
  75% subjects | 15 | 15
Statistical Analysis 1: Comparison: Placebo vs 700mg Leronlimab; Test type: Superiority; p = 0.4138, Likelihood test-Cox Prop. hazards model; Stratification factors: Baseline NEWS Total score and Age; Hazard Ratio (HR) = 0.781, 95% CI 2-sided [0.43 to 1.41]

3. Secondary Outcome: Incidence of Hospitalization
Description: Number of patients requiring hospitalization
Time Frame: From visit 2 (day 0) through day 14 (in days)
Population: MITT
Measure: Number; unit: participants
Arm/Group | Placebo | 700mg Leronlimab
Number analyzed (Participants) | 28 | 56
participants
  None | 11 | 22
  1 time | 14 | 33
  2 times | 3 | 1

4. Secondary Outcome: Duration (Days) of Hospitalization
Description: Duration of hospitalization in days
Time Frame: Total duration of hospitalization between visit 2 (day 0) in days and end of treatment
Population: MITT
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo | 700mg Leronlimab
Number analyzed (Participants) | 28 | 56
days | 2.0 (3.19) | 2.1 (3.83)

5. Secondary Outcome: Incidence of Mechanical Ventilation
Description: Incidence of mechanical ventilation supply
Time Frame: Total duration of mechanical ventilation since visit 2 (day 0) (days)
Population: MITT
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 700mg Leronlimab
Number analyzed (Participants) | 28 | 56
Participants
  None | 27 | 55
  1 Time | 1 | 1

6. Secondary Outcome: Duration of Mechanical Ventilation Supply
Description: Duration (days) of mechanical ventilation supply
Time Frame: Duration of mechanical ventilation since visit 2 (day 0) (days
Population: MITT
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo | 700mg Leronlimab
Number analyzed (Participants) | 28 | 56
days | 0.4 (1.96) | 0.2 (1.00)

7. Secondary Outcome: Incidence of Oxygen Use
Description: Incidence of oxygen use over course of treatment
Time Frame: Use of oxygen since visit 2 (day 0) to end of treatment
Population: MITT
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 700mg Leronlimab
Number analyzed (Participants) | 28 | 56
Participants
  None | 22 | 47
  One time | 5 | 6
  Two times | 1 | 2
  Three times | 0 | 1

8. Secondary Outcome: Duration of Oxygen Use
Description: Duration of oxygen use in days
Time Frame: Total duration of oxygen use since visit 2 (day 0) to EOT (day 14) (days)
Population: MITT
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo | 700mg Leronlimab
Number analyzed (Participants) | 28 | 56
days | 0.8 (2.81) | 0.9 (2.98)

9. Secondary Outcome: Mortality at Day 14
Description: Incidence of mortality at day 14
Time Frame: Mortality at EOT (day 14)
Population: MITT
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 700mg Leronlimab
Number analyzed (Participants) | 28 | 56
Participants | 0 | 0

10. Secondary Outcome: Time to Return to Normal Activity
Description: Time to return to normal activity from initiation of study treatment defined as duration from date of first exposure to treatment to the first occurrence of ordinal scale equals "not hospitalized, no limitations of activities"
Time Frame: Date of first exposure to treatment to the first occurrence of ordinal scale equals "not hospitalized, no limitations of activities"
Population: MITT
Measure: Number; unit: days
Arm/Group | Placebo | 700mg Leronlimab
Number analyzed (Participants) | 28 | 56
days
  25th percentile pts return to normal | 4.0 | 5.0
  50th percentile pts return to normal | 8.0 | 8.0
  75th percentile pts return to normal | 9.0 | 15.0

11. Secondary Outcome: Change From Baseline in National Early Warning Score 2 (NEWS2) to Day 3, 7 and 14
Description: NEWS2 is an assessment based on 7 clinical parameters (respiration rate, oxygen saturation, any supplemental oxygen, temperature, systolic blood pressure, heart rate, level of consciousness) developed by the Royal College of Physicians (https://www.rcplondon.ac.uk/projects/outputs/national-early-warning-score-news-2). Respiratory rate (bpm) scores 0-3; Sp02 (on room air or suppl) scores 0-3; SpO2 (hypercapnic resp failure) scores 0-3; room air or supplemental O2 scores 0 (room) or 2 (suppl); temperature - scores 0-3; systolic BP scores 0-3; pulse (bpm) scores 0-3; consciousness - alert (score 0) vs. new onset confusion (score 3). The total possible score ranges from 0 to 20. The higher the score the greater the clinical risk. Higher scores indicate the need for escalation, medical review and possible clinical intervention and more intensive monitoring.
  Change shown is positive or negative from baseline, with a negative number indicating improvement (i.e., a decrease in total score).
Time Frame: Baseline to Day 3, 7 and 14
Population: MITT
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | 700mg Leronlimab
Number analyzed (Participants) | 28 | 56
score on a scale
  Change from Baseline to Day 3 | 0.0 (0.87) | -0.3 (1.67)
  Change from Baseline to Day 7 | -0.2 (1.27) | -0.3 (2.24)
  Change from Baseline to Day 14 | -0.2 (1.06) | -0.4 (2.42)

12. Secondary Outcome: Mean Change in Percent Oxygen Saturation From Baseline to Days 3, 7 and 14
Description: Mean change in percent oxygen saturation from baseline to Days 3, 7 and 14 for patients with paired values
Time Frame: Mean change in percent oxygen saturation from baseline to Days 3, 7 and 14
Population: MITT
Measure: Mean (Standard Deviation); unit: Mean change in % O2 sat
Arm/Group | Placebo | 700mg Leronlimab
Number analyzed (Participants) | 28 | 56
Mean change in % O2 sat
  Mean change from Baseline to Day 3 of percent oxygen saturation | 0.3 (1.91) | -0.1 (2.0)
  Mean change from Baseline to Day 7 of percent oxygen saturation | 0.4 (2.08) | 0.00 (2.30)
  Mean change from Baseline to Day 14 of percent oxygen saturation | 0.6 (1.73) | 0.3 (2.39)

13. Secondary Outcome: Change From Baseline in the Patient's Health Status on a 7-category Ordinal Scale on Days 3, 7 and 14
Description: A 7-category ordinal scale of patient health status ranges from: 1) Death; 2) Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO); 3) Hospitalized, on non-invasive ventilation or high flow oxygen devices; 4) Hospitalized, requiring supplemental oxygen; 5) Hospitalized, not requiring supplemental oxygen; 6) Not hospitalized, limitation on activities; 7) Not hospitalized, no limitations on activities.
  Lower scores mean a worse outcome.
Time Frame: Assessments performed Day 0 (first treatment is Visit 2, day 0), Visit 3 (3+/- 1 day after first treatment) Visit 4 (second treatment, 7+/- 1 day from V2, day7) and end of treatment (7+/- 1 day from V4, day 14)
Population: MITT
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | 700mg Leronlimab
Number analyzed (Participants) | 28 | 56
units on a scale
  Mean change from baseline at day 3 | 0.4 (0.80) | 0.5 (0.75)
  Mean change from baseline at day 7 | 1.1 (0.78) | 0.7 (0.99)
  Mean change from baseline at day 14 | 1.2 (0.75) | 1.0 (1.13)

14. Other Pre Specified Outcome: Change in Size of Lesion Area by Chest Radiograph or CT
Description: Change in size of lesion area by chest radiograph or CT - exploratory endpoint
Time Frame: Day 14
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Change From Baseline in Serum Cytokine and Chemokine Levels
Description: Change from baseline in serum cytokine and chemokine levels at day 3, day 7 and day 14
Time Frame: Days 3, 7, and 14
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Change From Baseline in CCR5 Receptor Occupancy Levels for Tregs and Macrophages
Description: Change from baseline in CCR5 receptor occupancy levels for Tregs and macrophages at day3, day 7 and day 14
Time Frame: Days 3, 7, and 14
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Change From Baseline in CD3+, CD4+ and CD8+ T Cell Count
Description: Change from baseline in CD3+, CD4+ and CD8+ T cell count at day 3, day 7 and day 14
Time Frame: Days 3, 7, and 14
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Study drug was administered at Visit 2 (day 0) and visit 4 (day 7). Adverse events were assessed during the course of treatment and during the follow up period i.e., 2 weeks (visit 6) and 4 weeks (visit 7) after end of treatment. Therefore adverse events were assessed over a period of 5 weeks (visit 2 to visit 7).
Arm/Group | Placebo | 700mg Leronlimab
All-Cause Mortality (participants affected / at risk) | 0/28 | 1/56
Serious Adverse Events (participants affected / at risk) | 6/28 | 5/56
Other Adverse Events (participants affected / at risk) | 12/28 | 7/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=28) | 700mg Leronlimab (N=56)
Atrial Fibrillation (Cardiac disorders) | 1 | 0
Mitral Valve Incompetence (Cardiac disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 0
Chest Pain (General disorders) | 2 | 0
Death (General disorders) | 0 | 1
Swelling face (General disorders) | 1 | 0
Liver Abcess (Infections and infestations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Arterial occlusive disease (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=28) | 700mg Leronlimab (N=56)
Fatigue (General disorders) | 2 | 1
C-reactive protein increased (Investigations) | 1 | 3
Pneumonia (Infections and infestations) | 2 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-03-30): https://cdn.clinicaltrials.gov/large-docs/51/NCT04343651/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-26): https://cdn.clinicaltrials.gov/large-docs/51/NCT04343651/SAP_001.pdf